CLINICAL TRIAL: NCT04735367
Title: Retrospective, Multicenter, Observational Study to Evaluate Overall Survival in Japanese Patients With HR+/HER2- Advanced Breast Cancer Treated With Palbociclib Plus Letrozole
Brief Title: Study to Evaluate Overall Survival in Japanese Patients With HR+/HER2- Advanced Breast Cancer Treated With Palbociclib Plus Letrozole
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481154; NCT04735367 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: retrospective; multicenter; observational study; Japan; HR+/HER2- advanced breast cancer; palbociclib; overall survival
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: palbociclib plus letrozole — palbociclib plus letrozole

SUMMARY:
This is a retrospective, multicenter, observational study in Japan. The primary objective is to evaluate overall survival (OS) in Japanese patients with HR+/HER2- advanced breast cancer who have been treated with palbociclib plus letrozole. This observational study was planned as follow-up study of Japanese phase 2 study of palbociclib (NCT01684215, phase 2 portion of A5481010 study).

ELIGIBILITY:
Inclusion Criteria:

1. Participated, treated with palbociclib plus letrozole in J-Ph2, and was under follow-up for survival at the study completion of J-Ph2.
2. For patients who are still alive and have routine visits to the study site, evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study. For patients who are still alive and had been transferred to another hospital, evidence that the patient has been informed of all pertinent aspects of the study and oral or written informed consent is obtained. For patients who had already passed away, the conduct of this study will be disclosed, and the patients' legally acceptable representatives will be guaranteed an opportunity to refuse data collection for the patients in accordance with the Ethical Guidelines for Medical and Health Research Involving Human Subjects

Exclusion Criteria:

1. There are no exclusion criteria for this study.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who participated, treated with palbociclib plus letrozole, and under follow-up for survival in J-Ph2
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- Japan (13):
  - Chiba cancer center, Chiba, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Saitama Cancer Center, Kita-adachi-gun, Saitama
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hakuaikai Medical Corporation Sagara Hospital, Kagoshima
  - Kumamoto Shinto General Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Aichi Cancer Center, Nagoya
  - National Hospital Organization - Osaka National Hospital - Institute For Clinical Research, Osaka

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Takahashi M, Yasojima H, Osako T, Inoue K, Kawashima M, Maeda H, Ito M, Sagara Y, Yonemori K, Hattori M, Yamamoto N, Muramatsu Y, Matsui A, Masuda N. Overall survival and subsequent therapy patterns in Japanese patients with ER+/HER2- advanced breast cancer treated with palbociclib plus letrozole in the first-line setting: a final analysis. Breast Cancer. 2025 Nov;32(6):1482-1490. doi: 10.1007/s12282-025-01760-0. Epub 2025 Aug 21. PMID 40841781
- [Derived] Takahashi M, Osako T, Yasojima H, Inoue K, Kawashima M, Maeda H, Ichikawa A, Muramatsu Y, Masuda N. Overall survival in Japanese patients with ER+/HER2- advanced breast cancer treated with first-line palbociclib plus letrozole. Breast Cancer. 2024 Jan;31(1):53-62. doi: 10.1007/s12282-023-01511-z. Epub 2023 Oct 26. PMID 37882974
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481154

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data was collected from participants who were treated with palbociclib plus letrozole in Japanese Phase 2 study A5481010 (NCT01684215). Data was collected retrospectively from individual participant medical records for participants under survival follow up at the time of completion of study A5481010 and for participants who died or refused follow-up in study A5481010, data collected in Phase 2 study was used for analysis.
Groups:
- Palbociclib+ Letrozole: Participants with hormone receptor positive/human epidermal growth factor receptor 2 negative (HR+/HER2-) advanced breast cancer who were treated with palbociclib plus letrozole in study A5481010 (NCT01684215).
Period: Overall Study
Arm/Group | Palbociclib+ Letrozole
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis set included participants who were enrolled in Japanese Phase 2 (J-Ph2) study and received the investigational product, excluding surviving participants who did not give written or oral consent.
Groups:
- Palbociclib+ Letrozole: Participants with HR+/HER2- advanced breast cancer who were treated with palbociclib plus letrozole in study A5481010 (NCT01684215).
Arm/Group | Palbociclib+ Letrozole
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose of the investigational product in Japanese Phase 2 study (A5481010) to the date of any-cause death. In the absence of confirmation of death, survival time was censored to last date the participant was known to be alive. Kaplan-Meier method was used for analysis.
Time Frame: From the date of the first dose of the treatment in study A5481010 to the date of any-cause death or censoring date (maximum of 103.16 months of follow-up); data collected and observed retrospectively over 32 months in A5481154 study
Population: Analysis set included participants who were enrolled in J-Ph2 and received the investigational product excluding surviving participants who did not give written or oral consent.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib+ Letrozole
Number analyzed (Participants) | 42
Months | 85.42 [64.26 to NA] — Upper limit of 95% confidence interval (CI) could not be estimated because of insufficient number of participants with events.

2. Secondary Outcome: Percentage of Participants According to Types and Line of Subsequent Treatment
Description: Participants were classified based on types of subsequent treatment and by line of subsequent treatment. Subsequent treatments included: endocrine therapy-based, chemotherapy-based and others (Investigational drug + Endocrine therapy/Chemotherapy).
Time Frame: From start of subsequent treatment in study A5481010 until date of death, withdrawal of consent or end of study (maximum of 103.16 months of follow-up); data collected and observed retrospectively over 32 months in A5481154 study
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib+ Letrozole
Number analyzed (Participants) | 42
Percentage of participants
  Received First Subsequent Therapy | 81.0
  First Subsequent Therapy: Endocrine-based therapy | 69.0
  First Subsequent Therapy: Endocrine therapy + Chemotherapy | 0.0
  First Subsequent Therapy: Chemotherapy | 7.1
  First Subsequent Therapy: Other | 4.8
  Received Second Subsequent Therapy | 69.0
  Second Subsequent Therapy: Endocrine-based therapy | 40.5
  Second Subsequent Therapy: Endocrine therapy + Chemotherapy | 2.4
  Second Subsequent Therapy: Chemotherapy | 21.4
  Second Subsequent Therapy: Other | 4.8

3. Secondary Outcome: Duration of Subsequent Therapy by Line of Therapy
Description: Duration of subsequent therapy defined as time from the start date to the end date of each line of treatment among participants who received subsequent treatment. Kaplan-Meier method was used.
Time Frame: as for outcome 2
Population: Analysis set included participants who were enrolled in J-Ph2 and received the investigational product excluding surviving participants who did not give written or oral consent. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here "Number Analyzed" refers to the number of participants evaluable for the specified rows.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib+ Letrozole
Number analyzed (Participants) | 42
Months
  First Subsequent Therapy: number analyzed (Participants) | 34
  First Subsequent Therapy | 7.64 [3.91 to 9.00]
  Second Subsequent Therapy: number analyzed (Participants) | 29
  Second Subsequent Therapy | 6.01 [3.25 to 14.88]

ADVERSE EVENTS:
Time Frame: For all-cause mortality: From start of subsequent treatment in study A5481010 until date of death, withdrawal of consent or end of study (maximum of 103.16 months of follow-up); data collected and observed retrospectively over 32 months in study A5481154. Data for non-serious adverse events and serious adverse events (SAEs) were not collected and evaluated during the study; hence timeframe is not applicable for non-SAEs and SAEs.
Description: This observational retrospective study retrieved data from medical records and the data existed as unstructured data. In these data sources, individual participant data were not retrieved or validated. Hence adverse events were not assessed/collected.
Arm/Group | Palbociclib+ Letrozole
All-Cause Mortality (participants affected / at risk) | 20/42
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT04735367/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT04735367/SAP_001.pdf